CLINICAL TRIAL: NCT00440986
Title: Clinical Management of Hereditary Hemochromatosis: Phlebotomy vs. Erythrocytoapheresis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: San Filippo Neri General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMHHPE; HH1
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Hereditary Hemochromatosis
Keywords: Clinical Management; Phlebotomy; Eritrocytoapheresis
MeSH Terms: conditions — Hemochromatosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Eritrocytoapheresis

SUMMARY:
The purpose of study is to determine the best and durable choice of treatment between phlebotomy and eritrocytoapheresis in the medium- and long-term clinical management of HH

DETAILED DESCRIPTION:
Patients affected by Hereditary hemochromatosis need a completeinitial staging of disease, a correct clinical management, a good chance of treatment and long-term follow-up. Clinical manifestations at presentation and during follow-up may consistently vary according to diagnostic criteria, treatment options and follow-up durability, up to the interruption. So, 25 caucasian patients, 16 males and 6 females of age >18 yrs. have been consecutively diagnosed and randomly included into two arms of treatment, phlebotomy vs. eritrocytoapheresis, evaluating, at baseline and 6-12-18-24-36 months, the clinical status concerning liver, kidney, pancreas, heart, endocrine iron overload and function and final outcome related to therapeutic strategy, including the cost/effectiveness analysis

ELIGIBILITY:
Inclusion Criteria:

* Patiens newly diagnosed having Hereditary Hemochromatosis

Exclusion Criteria:

* Age < 18 yrs.
* Not obese (BMI <30)
* Not consuming alchol beverages,
* Not affected by systemic diseases and known hepatic viruses

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2003-04; Study Completion 2006-12

PRIMARY OUTCOMES:
To prospectively determine the best choice of tretment in HH
To evaluate the global outcome according to treatment choice

SECONDARY OUTCOMES:
To evaluate the outcome of specific clinical features according to treatment choice

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Equitani, M.D., Principal Investigator — San Filippo Neri General Hospital
Locations (1):
- Department of Transfusion Medicine-San Filippo Neri General Hospital, Rome, Italy

REFERENCES:
- [Background] Pietrangelo A. Hereditary hemochromatosis--a new look at an old disease. N Engl J Med. 2004 Jun 3;350(23):2383-97. doi: 10.1056/NEJMra031573. No abstract available. PMID 15175440
- [Derived] Equitani F, Fernandez-Real JM, Menichella G, Koch M, Calvani M, Nobili V, Mingrone G, Manco M. Bloodletting ameliorates insulin sensitivity and secretion in parallel to reducing liver iron in carriers of HFE gene mutations. Diabetes Care. 2008 Jan;31(1):3-8. doi: 10.2337/dc07-0939. Epub 2007 Oct 24. PMID 17959863